CLINICAL TRIAL: NCT07016945
Title: Reactions to Experiencing Distress (RED) Study
Brief Title: Reactions to Distress (RED) In Louisville, KY Study
Acronym: RED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: iRIS234741
Record Dates: First submitted 2025-06-02; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Threat Sensitivity
Keywords: attention bias; mindfulness; stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Main sample (Experimental): Participants are randomized to experimental and intervention conditions. They are either in: race stress/mindfulness, race stress/control audio, control stress/mindfulness, or control stress/control audio.
  Interventions: Behavioral: Stress and Mindfulness Intervention

INTERVENTIONS:
Behavioral: Stress and Mindfulness Intervention — Participants will be randomized to either the race-related stress condition or the non-race-related stress condition and the experimental group (7-minute pre-recorded audio file of a guided mindfulness practice) or the control group (7-minute pre-recorded neutral audio file). Thus there are four conditions total (RRS/Control Audio, RRS/Mindfulness Audio, Control Stress/Control Audio, Control Stress/Mindfulness Audio)

SUMMARY:
The goal of this study is to understand whether race-related stress can impact the way people direct their attention and what interventions may be helpful for attention.

DETAILED DESCRIPTION:
Race-related stress is a public health problem and a known predictor of severe psychological symptoms in Black Americans. Although there is a strong link between race-related stress and adverse mental health outcomes, limited research has examined the transdiagnostic mechanisms that explain how experiencing race-related stress contributes to psychological symptoms or what interventions might effectively target these mechanisms. The scientific premise of this study is that race-related stress may contribute to disproportionate allocation of attention toward threatening stimuli (i.e., attention bias to threat), a known predictor of stress-related symptoms. This attentional bias may be modifiable through a brief, culturally-informed mindfulness intervention.

Racial identity is hypothesized to be a key individual difference factor that influences the extent to which race-related stress affects attention bias to threat, as well as the degree to which a mindfulness intervention can mitigate these biases. The study will recruit 200 Black adults from the community who have experienced race-related stress to participate in a laboratory study targeting three specific aims:

To use eye-tracking methods to examine whether race-related stress (compared to non-race-related stress) leads to greater attention bias to threat;

To test whether a brief mindfulness meditation (compared to a neutral audio condition) reduces attention bias to threat;

To investigate whether racial identity moderates (a) the effect of the race-related stress manipulation on attention bias to threat and (b) the efficacy of the mindfulness intervention in reducing attention bias to threat.

This project includes a strong undergraduate training component designed to promote student engagement in psychological research and provide hands-on experience and comprehensive mentorship to support future research careers.

This research addresses critical gaps in the literature by investigating how race-related stress influences threat-related attentional processes, evaluating whether these processes can be altered by mindfulness-based strategies, and identifying for whom such interventions are most effective. The study utilizes a novel manipulation of race-related stress, an objective and theoretically grounded psychological mechanism (attention bias), precise assessment tools (eye-tracking), and an experimentally manipulated intervention (mindfulness), thereby addressing key limitations in existing research. Findings are expected to advance understanding of the psychological effects of racism and inform strategies to reduce mental health disparities among historically marginalized and underserved populations.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility for this study will include a positive response to the following questions: 1) Do you identify as Black or African American? 2) Have you ever in your lifetime personally experienced or witnessed another person experience any acts of racism or racial microaggressions? 3) Are you willing to complete a 1.5-hour study at the University of Louisville in the next 2 weeks? 4) Are you 18 or older?

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Free viewing task | 10 minutes
  Free Viewing Task. This is the outcome measure for both manipulations listed above. To assess attention bias to threat, we will use a free-viewing task in which participants are instructed to freely view a pair of images side by side across two blocks of 60 trials each. In Block 1, participants will view two types of image pairs: one threatening (i.e., angry face) and one neutral (i.e., neutral facial expression) or both neutral.
Affect | 5 minutes
  To ensure that the manipulations outlined above are having the intended effect (increase in NA/ decrease in PA after stress manipulation and the opposite after the mindfulness manipulation), participants will complete the 20-item PANAS after each manipulation. The items ask participants to indicate how they are feeling in the moment in terms of both negative affect (e.g., distressed, interested) and positive affect (e.g., strong, inspired) on a scale of 1 (very slightly or not at all) to 5 (very much). Scores are summed to create a total negative affect and positive affect score.

CONTACTS AND LOCATIONS:
Locations (1):
- Davidson Hall, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No
All relevant data are regularly uploaded to NIH NDA system.

DOCUMENTS (1):
  • Study Protocol (2025-06-02): https://cdn.clinicaltrials.gov/large-docs/45/NCT07016945/Prot_000.pdf